CLINICAL TRIAL: NCT03921801
Title: Improving Plantarflexor Muscle Function to Alleviate Decline in Mobility, Loss of Balance and Detrimental Knee Joint Loading in Older Adults
Brief Title: Effects of Improved Calf Muscle Function on Gait, Balance and Joint Loading in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Lauri Stenroth, Senior Researcher, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: LS_Plantarflex
Record Dates: First submitted 2018-12-10; First posted 2019-04-19 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee; Mobility Limitation; Accidental Fall
Keywords: Osteoarthritis; Knee; Achilles tendon; Triceps surae; Balance; Electromyography; Biofeedback; Strength training; Gait; Walking
MeSH Terms: conditions — Osteoarthritis, Knee; Mobility Limitation; Osteoarthritis | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Thirty older adults will be recruited and randomized into two groups. The other groups receive an intervention including strength training and gait retraining lasting 8 weeks while the other group receives only the gait retraining. Outcome measures are obtained before and after the intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait retraining (Active Comparator): 8-week intervention. Intervention includes weekly gait retraining sessions with real-time electromyography biofeedback.
  Interventions: Other: Gait retraining
- Gait retraining + strength training (Experimental): 8-week intervention. Intervention includes weekly gait retraining sessions with real-time electromyography biofeedback and home-based strength training session for plantarflexor muscles three times per week.
  Interventions: Other: Gait retraining + strength training

INTERVENTIONS:
Other: Gait retraining — Gait retraining using real-time electromyography biofeedback performed once per week for eight weeks.
  During the gait retraining session the participant is walking on a treadmill while receiving information on calf muscle activation. A single session includes five bouts of walking each lasting for 5 minutes. During the first bout, the participant is receiving feedback (visual and auditive) on soleus muscle activation with the aim to increase it by 20% from their normal walking. During the second bout, the participant is receiving feedback (visual and auditive) on medial gastrocnemius muscle activation with the aim to decrease it by 20% from their normal walking. During the last three bouts, the participant is receiving feedback (visual and auditive) on the soleus to medial gastrocnemius muscle activation ratio with the aim to increase it by 20% from their normal walking. If hitting the target, the aim is increased by 5% for the subsequent bout.
  Arms: Gait retraining
Other: Gait retraining + strength training — Gait retraining using real-time electromyography biofeedback performed once per week and home-based calf muscle strength training performed three times per week for eight weeks.
  The gait retraining is identical to the one intervention described for the intervention group "Gait retraining".
  The strength training is performed three times per week except for the first week in which it is performed two times. The session contained a warm-up (3x10 repetitions of two-legged heel raises) and maximal isometric calf muscle contractions. The maximal contractions are performed using a custom device with the ankle in dorsiflexion and the knee flexed by 100-120 degrees. Three sets of 10 repetitions (3-second contraction and 3-second rest) are performed with both legs and with maximal effort and 1-minute rest between the sets.
  Arms: Gait retraining + strength training

SUMMARY:
This study investigates the role of calf muscle function in gait performance, balance and knee joint loading.

Previous studies have linked age-related loss of calf muscle function with impairments in gait performance and balance, and increased loading of the areas of the knee joint that are susceptible to the development of osteoarthritis. In this study, an exercise intervention targeting structural and neural aspects of impaired calf muscle function with ageing is utilized. The intervention lasts 8 weeks and includes either biofeedback training using electromyography to alter muscle activation patterns or a combination of biofeedback training and strength training for the calf muscle to modify calf function during walking. The study will test whether the intervention improves walking speed, reduces the metabolic cost of walking, improves standing balance and reduces knee joint loading.

ELIGIBILITY:
Inclusion Criteria:

* age between 65 and 75

Exclusion Criteria:

* dependent living status
* not able to walk without an assistive device or for 30 min without stopping
* diagnosed neurological disease or joint disorder and pain during walking
* surgery on lower extremities
* current musculoskeletal injury
* previous cardiovascular event or symptoms during exercise (acute ECG change, coronary disease, symptomatic arrhythmia, symptomatic coronary stenosis, heart failure, myocarditis, pericarditis, pulmonary embolism, pulmonary infarct, artery bulge or rupture risk)
* body mass index <18 or >35 kg/m2
* contraindications for magnetic resonance imaging
* Mini Mental State Examination score of 23 points and lower

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Change from baseline in knee joint loading | within 1 weeks after intervention
  Change in tibiofemoral compressive loading during walking estimated using musculoskeletal modeling and simulation. Loading is calculated separately for medial and lateral compartments of the tibiofemoral joint.

SECONDARY OUTCOMES:
Change from baseline in energy cost of walking | within 1 weeks after intervention
  Assessed using indirect calorimetry.
Change from baseline in standing balance | within 1 weeks after intervention
  Sway during standing measured using a force plate with eyes open and closed
Change from baseline in Achilles tendon stiffness | within 1 weeks after intervention
  Achilles tendon stiffness evaluated using combination of ultrasonography, motion analysis and force measurements.
Change from baseline in gait kinematics | within 1 weeks after intervention
  Time series of lower limb joint angles during walking stride assessed using motion capture system and inverse kinematics.
Change from baseline in joint moments during walking | within 1 weeks after intervention
  Time series of lower limb joint moments during walking stride assessed using inverse dynamics based on motion capture system and instrumented treadmill data.
Change from baseline in joint powers during walking | within 1 weeks after intervention
  Time series of lower limb joint powers during walking stride assessed using inverse dynamics based on motion capture system and instrumented treadmill data.
Change from baseline in distribution of joint work during walking | within 1 weeks after intervention
  Distribution of total positive lower limb work between the joints during walking assessed using inverse dynamics based on motion capture system and instrumented treadmill data.
Change from baseline in muscle-tendon function during walking | within 1 weeks after intervention
  Muscle fascicle kinematics measured using dynamics ultrasonography during walking.
Change from baseline in soleus to gastrocnemius muscle activation ratio | within 1 weeks after intervention
  Relative activation of soleus to medial gastrocnemius measured using electromyography.
Change from baseline in walking speed | within 1 weeks after intervention
  Preferred and maximal walking speed.
Change from baseline in muscle strength | within 1 weeks after intervention
  Maximal isometric muscle strength in ankle plantarflexion and knee extension and flexion.

OTHER OUTCOMES:
Change from baseline in triceps surae fascicle lengths | within 1 weeks after intervention
  Soleus and gastrocnemius muscle fascicle length assessed using ultrasound imaging.
Change from baseline in triceps surae fascicle pennation angle | within 1 weeks after intervention
  Soleus and gastrocnemius muscle pennation angle assessed using ultrasound imaging.
Change from baseline in triceps surae muscle volume | within 1 weeks after intervention
  Soleus and gastrocnemius muscle volume estimated with combination of ultrasound and magnetic resonance imaging.
Change from baseline in Achilles tendon cross-sectional area | within 1 weeks after intervention
  Achilles tendon cross-sectional area assessed using magnetic resonance imaging.
Change from baseline in dynamics balance control | within 1 weeks after intervention
  Perturbed standing balance test with measurement of center of pressure trajectory
Change from baseline in triceps surae muscle activity in response to balance perturbation | within 1 weeks after intervention
  Perturbed standing balance test with measurement of triceps surae muscle activities.

CONTACTS AND LOCATIONS:
Overall Officials: Lauri Stenroth, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: Yes
Data obtained during the study will be shared with other researcher after the results have been published. Details of the data will be updated later.
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication
Access Criteria: At request from the principal investigator.